CLINICAL TRIAL: NCT05547139
Title: Impact of Extended CPAP Utilization on Bronchopulmonary Dysplasia in Extremely Premature Infants: A Pilot Randomized Control Trial
Brief Title: Impact of Extended CPAP on Bronchopulmonary Dysplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 605186
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Bronchopulmonary Dysplasia; Prematurity
Keywords: Bronchopulmonary dysplasia; Prematurity; High flow nasal cannula; Continuous positive airway pressure; NICU
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Intervention Model Description: Infants will be randomized to the usual care group or the protocol care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (No Intervention): Infants randomized to this group will receive the present standard of care for weaning respiratory support. This means the attending provider will decide when each infant is ready to be changed from CPAP to nasal cannula and the nasal cannula will be weaned according to an existing unit protocol.
- Protocol care group (Active Comparator): Infants randomized to this group will remain on CPAP until they are at least 32 weeks corrected gestational age or 1250g. At that point, if they meet a set of criteria, they will be transitioned to either 2L nasal cannula if they require supplemental oxygen or room air.
  Interventions: Other: Protocolized weaning of respiratory support

INTERVENTIONS:
Other: Protocolized weaning of respiratory support — The protocolized weaning aims to keep babies on CPAP for a longer period of time and will measure how long it takes babies to wean to 2L nasal cannula support or come off all support (room air, RA).
  Arms: Protocol care group

SUMMARY:
The purpose of this pilot study is to compare if keeping infants on CPAP (continuous positive airway pressure) support for an extended period of time until they are 32 weeks corrected gestational age or 1250 grams (approximately 2 pounds and 12 ounces) will decrease their degree of lung disease as compared to weaning their respiratory support to HFNC (high flow nasal cannula).

DETAILED DESCRIPTION:
There are two ways to help premature babies breathe. Both HFNC and CPAP are commonly used in our NICU. CPAP, which helps your baby breathe without a tube in their windpipe (intubation or ventilator), delivers oxygen and air by pressure through either small prongs in the nose or a nose mask, keeping your baby's airways open. HFNC provides heated and humidified oxygen and air by small prongs in the nose that does not use high pressure to the airways. Our goals are to reduce long term complications such as lung disease of prematurity, also called Bronchopulmonary Dysplasia (BPD). BPD causes "lung damage/scarring, need for a ventilator or oxygen, brain/neurological impairment etc. In recent years, HFNC has become a common choice for care. There is no clear agreement in previous research which way may be best to reduce BPD.

ELIGIBILITY:
Inclusion Criteria:

* babies born at <30 weeks' gestation
* babies who are extubated to non-invasive ventilation by 32 weeks postmenstrual age

Exclusion Criteria:

* babies born at <30 weeks' gestation
* requiring less than 2L NC at birth or
* those who are extubated after 32.0 weeks' postmenstrual age
* congenital anomalies
* skeletal disorders
* neuromuscular disorders
* genetic syndromes

Ages: 22 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Time to reach 2L NC or room air | up to 3 months
  The primary outcome is time (in days) to reach 2L nasal cannula or room air

SECONDARY OUTCOMES:
Compliance to protocol and balancing measures | up to 3 months
  compliance to intervention, medical team attitude towards intervention, death, pneumothorax after extubation, septal breakdown, necrotizing enterocolitis (NEC), number of failed wean off respiratory support attempts, duration of noninvasive respiratory support, failure to maintain non-invasive support, duration of Fi02 requirement >21%, need for systemic steroids, time to full enteral feeds, time to initiation of PO feeds, time to >75% PO feeds, length of stay, and growth velocity at discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Z Kovatis, MD, Principal Investigator — Christiana Care Health Services, Inc; Anastasiya Latushko, Principal Investigator — Christiana Care Health Services, Inc
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No